CLINICAL TRIAL: NCT06651177
Title: NIDA CTN-0152: Evaluation of Tirzepatide as an Adjunct to Buprenorphine for the Treatment of Opioid Use Disorder: A Pragmatic, Multi-site, Double-blind, Randomized, Placebo-controlled Trial (TAB)
Brief Title: Evaluation of Tirzepatide as an Adjunct to Buprenorphine for the Treatment of Opioid Use Disorder
Acronym: TAB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: T. John Winhusen, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-1003; UG1DA013732 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Opioid Use Disorder, Moderate; Opioid Use Disorder, Severe
Keywords: tirzepatide; opioid; opioid use disorder; buprenorphine; GLP-1
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): The tirzepatide pen is a pre-filled, disposable, injection device designed for subcutaneous administration. Each pen is pre-filled with a single dose of tirzepatide and is available in six doses: 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg, and 15 mg/0.5 mL. An unblinded study MC (UMC) will administer the once-weekly SQ dose of tirzepatide. Consistent with tirzepatide's prescribing guidelines, participants will be initiated at a once-weekly SQ dose of 2.5 mg/week with a dose increase to 5mg/week at week 5. Consistent with tirzepatide's prescribing information, once the participant has received 5 mg/week for 4 weeks they are eligible for a dose increase if needed.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Saline administered subcutaneously with a syringe will be used as the placebo for the trial. The placebo which will be administered by a study UMC. The process for deciding on "dose increases" will be the same for placebo and tirzepatide.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — The tirzepatide pen is a pre-filled, disposable, injection device designed for subcutaneous administration. Each pen is pre-filled with a single dose of tirzepatide and is available in six doses: 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg, and 15 mg/0.5 mL. A UMC will administer the once-weekly SQ dose of tirzepatide. Consistent with tirzepatide's prescribing guidelines, participants will be initiated at a once-weekly SQ dose of 2.5 mg/week with a dose increase to 5mg/week at week 5. Consistent with tirzepatide's prescribing information, once the participant has received 5 mg/week for 4 weeks they are eligible for a dose increase if needed
  Other Names: Mounjaro; Zepbound
  Arms: Tirzepatide
Other: Placebo — Saline administered subcutaneously with a syringe will be used as the placebo for the trial. The placebo which will be administered by a study UMC. The process for deciding on "dose increases" will be the same for placebo and tirzepatide.
  Arms: Placebo

SUMMARY:
The primary objective of this research study is to evaluate the effect of tirzepatide, relative to placebo, as an adjunct to BUP on retention, substance use, and sleep outcomes in individuals with OUD.

DETAILED DESCRIPTION:
This is a Phase 2, pragmatic, multi-site, double-blind, randomized, placebo-controlled, intent-to-treat trial. The selection of placebo as the comparator is considered the gold standard for medication trials. Eligible participants will be randomized in a 1:1 ratio to tirzepatide or placebo, balancing on site and buprenorphine (BUP) formulation (transmucosal vs extended-release).

Participants will receive tirzepatide or placebo based on randomized assignment, with "dose escalation" of placebo following the schedule for tirzepatide and tirzepatide dosing being consistent with prescribing guidelines. Participants will be administered a subcutaneous (SQ) study medication injection weekly and attend weekly research visits through 26 weeks post-randomization with longer research visits at 1, 3, and 6 months post-randomization. A follow-up visit for final safety measures will be completed at week 30, which takes into account tirzepatide's long half-life.

Duration of participation will be approximately 31 weeks for study participants. Participants will be administered study medication and attend weekly research visits through 6 months post-randomization with longer research visits at 1-, 3-, and 6-months post-randomization. Participants will be provided with a Fitbit to measure sleep. BUP is not a study medication; participants will receive BUP through their clinical provider. A follow-up visit for final safety measures will be completed at week 30.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age;
2. Must have moderate to severe OUD;
3. Must, at the time of randomization, be newly initiated on BUP (i.e., within 7 to 28 days) during the current treatment episode, be taking ≥ the recommended target dose for transmucosal BUP (or equivalent for extended-release), and have documentation of receiving BUP, including dose and the start date of the current treatment episode, from their BUP provider;
4. Must be willing to be randomized to tirzepatide or placebo and to comply with study procedures, including weekly visits for 6 months;
5. Must be able to understand the study, and having understood, provide written informed consent in English;
6. Must not be breastfeeding; if of child bearing potential, must test negative on the study-administered pregnancy test(s), and if of childbearing potential and engaging /planning to engage in sexual intercourse must agree to effective contraception for the duration of the trial through 30 days after the trial; effective contraception is defined as using: a) birth control injection, an intrauterine device, or implant; or b) two birth control methods - for example birth control pills with a barrier method (e.g., condoms, etc.).

   * If ever of childbearing potential, a participant is considered to not be of childbearing potential for the study if they are:

     1. infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, tubal implants, or tubal ligation), congenital anomaly such as Mullerian agenesis; are
     2. post-menopausal defined as ≥ 55 years old not on hormone therapy, who has had at least 12 months of spontaneous amenorrhea;
     3. ≥ 55 years old with a diagnosis of menopause prior to starting hormone replacement therapy; or
     4. ≥ 40 years old with an intact uterus, not on hormone therapy, who has cessation of menses for at least 1 year without an alternative medical cause, AND a follicle-stimulating hormone ≥ 40 mIU/mL; participants in this category must test negative on the study-administered pregnancy test(s).

Exclusion Criteria:

1. have a history of type 1 or type 2 diabetes mellitus (other than pregnancy-related diabetes);
2. have a BMI <25.0;
3. have any of the following cardiovascular conditions within 90 days prior to signing consent: acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or hospitalization due to congestive heart failure (CHF);
4. have a known history of chronic or acute pancreatitis, gallbladder disease, gastroparesis, gastric emptying abnormality, gastroesophageal reflux disease, or other severe gastrointestinal disease;
5. have a personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2);
6. have previously taken tirzepatide, have taken any GLP-1 analogue within the 6 months before consent, or have a known history of prior hypersensitivity reaction to any GLP-1 analogue;
7. have renal impairment defined as an estimated glomerular filtration rate (eGFR) value of < 15 mL/min/1.73 m2 or requiring dialysis;
8. have a current, or within the 30 days prior to signing consent, use of, or plan to start during the course of the trial:

   1. medications with glucose lowering properties: GLP-1 analogs, sulfonylurea, insulin, metformin, thiazolidinediones, dipeptidyl peptidase-4 (DPP-IV) inhibitors, sodium-glucose cotransporter-2 (SGLT-2) inhibitors;
   2. systemic steroids including prednisone, hydrocortisone, dexamethasone;
9. have a history of suicide attempts or significant active suicidal ideation as assessed by a qualified study clinician;
10. have a psychiatric or medical condition that, in the judgment of the site medical clinician (BMC or UMC), would make study participation unsafe or which would make treatment compliance difficult;
11. have current status as a prisoner OR be currently in jail, prison, or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that, in the judgement of the site investigator, could prevent participation in the study or in any study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
6-month medication for opioid use disorder (MOUD) retention rate - Timeline Follow-Back (TLFB) | 6 months
  MOUD is defined as buprenorphine (BUP) or methadone. The receipt of MOUD will be assessed by self-report collected through a TLFB procedure.
6-month medication for opioid use disorder (MOUD) retention rate - Urine Drug Screen (UDS) | 6 months
  MOUD is defined as BUP. This will be measured by UDS results for BUP.

SECONDARY OUTCOMES:
Proportion of illicit opioid-negative urine samples during the 6-month active treatment phase | 6 Months
  A rapid Urine Drug Screen (UDS)UDS system will be used to analyze the urine samples. Urine samples will be tested for: buprenorphine/ norbuprenorphine and fentanyl.
Proportion of urine samples negative for other substances of abuse during the 6-month active treatment phase | 6 months
  Nicotine abstinence will be assessed with cotinine, alcohol abstinence will be assessed with ethyl glucuronide, and drug abstinence will be assessed based on the other substances (other than buprenorphine/ norbuprenorphine) assessed for by the UDS system.
Substance Use Days | 6 months
  Days of illicit-opioid, other drug, alcohol, and nicotine use during the 26 week active treatment phase will be assessed with the Timeline Follow-back (TLFB).
Days of Substance Bingeing | 6 months
  Days of bingeing of illicit opioids and/or other drugs during the 26 week active treatment phase will be assessed with the Timeline Follow-back (TLFB).
Opioid Cravings | 6 months
  Craving will be assessed with the Opioid Craving Scale, which was utilized in CTN-0030 and shown to have predictive validity. The total score is calculated by averaging the scores from three visual analogue scales which assess craving, cue-induced craving, and likelihood of using.
Opioid Withdrawal Symptoms | 6 months
  The Short Opiate Withdrawal Scale (SOWS)-Gossop will be used to measure opioid withdrawal symptoms. The SOWS-Gossop, which is a self-administered scale that includes 10 items, rated on a scale of 0 (none) to 3 (severe), is a validated instrument with good reliability.
The Modified Patient-Reported Outcomes Measurement Information System (PROMIS)-based Opioid Use Monitor | 6 months
  The PROMIS-based Opioid Use Monitor (OUM) was adapted from the PROMIS substance use measure by replacing "drugs" with "opioids" and changing the timeframe from the past 3 months to the past 2 weeks. For the present trial, a modified version of the OUM (M-OUM) will be used as an outcome measure and for use in determining whether a dose increase is needed. The M-OUM includes seven items that are each rated on a 0-4-point scale ("0-never" to "4-almost always") yielding a total score of 0-28.
Treatment Effectiveness | 6 months
  Treatment Effectiveness will be measured by the Treatment Effectiveness Assessment (TEA). The TEA is a patient-oriented instrument that assesses the participant's perceived improvements in substance use, health, ability to fulfill adult obligations, and to be a good community member. The TEA includes four items, each rated on a 1-10-point scale (from none to much better) yielding a total score of 4-40.
Non-Opioid Drug and Alcohol Craving | 6 months
  Non-Opioid Drug and Alcohol Craving will be measured by the Non-Opioid Drug and Alcohol Craving Scale. The 3-item craving scale, which assesses craving for drugs and alcohol, will be modified to ask about substances other than opioids.
Self-reported control of opioid/stimulant use and craving - | 6 months
  The PROMIS-based Opioid Use Monitor (OUM) was adapted from the PROMIS substance use measure by replacing "drugs" with "opioids" and changing the timeframe from the past 3 months to the past 2 weeks. A modified version of the OUM (M-OUM) will be used as an outcome measure and for use in helping to determine whether a dose increase should be offered.
Sleep Quality - Fitbit Charge 6™ (FBC-6) | 6 months
  An objective measure of the impact of tirzepatide, relative to placebo, on sleep will be obtained using the Fitbit Charge 6™ (FBC-6). A comparison of an earlier version of the device (Fitbit Charge 4™) to polysomnography found no significant differences in the measures of total sleep time and waking after sleep onset. Each participant will be provided with a Fitbit Charge 6™ when they are deemed eligible for randomization and asked to wear it every night (or whenever they have their longer period of intended sleep) through the final study visit. Data from the Fitbit Charge 6™ will be downloaded at the weekly research visits. Total sleep time is the main outcome of interest.
Sleep Quality - The Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Participant perceived sleep quality will be assessed using the PSQI, which is a relatively brief, validated instrument that measures sleep quality.

OTHER OUTCOMES:
Metabolic-related outcomes - A1C | 6 months
  Blood samples to assess A1C will be obtained at baseline, month 3, and month 6. Mean change in A1C (%) is the outcome of interest.
Metabolic-related outcomes - Body Mass Index (BMI) | 6 months
  Height will be measured at screening/baseline and weight will be measured. Body mass index (BMI) will be calculated with mean change in BMI (kg/m2) as the outcome of interest.
Metabolic-related outcomes - Weight | 6 months
  Weight will be measured. Mean change in weight (kg) is the outcome of interest.
Metabolic-related outcomes - % Weight loss | 6 months
  Weight will be measured. Proportion of weight loss (kg) is the outcome of interest.

CONTACTS AND LOCATIONS:
Overall Officials: T. John Winhusen, PhD., Principal Investigator — University of Cincinnati
Locations (10):
- United States (10):
  - Tarzana Treatment Centers, Tarzana, California
  - Gateway Community Services, Jacksonville, Florida
  - IBIS Behavioral Health, Tampa, Florida
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - The Gibson Center for Behavioral Change, Cape Girardeau, Missouri
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Marshall Health, Huntington, West Virginia
  - Healthy Minds/Chestnut Ridge, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data gathered from case report forms.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 11, 2028 (anticipated)
Access Criteria: Primary data for this study will be available to the public in the NIDA data repository, per NIDA CTN policy. For more details on data sharing please visit https://datashare.nida.nih.gov/.
URL: https://datashare.nida.nih.gov/